CLINICAL TRIAL: NCT04470466
Title: Short Pulse and Q-switched ND-YAG Laser With Topical Carbon Versus Fractional CO2 Laser in Treatment of Enlarged Facial Pores: A Split-face Comparative Study
Brief Title: Short Pulse and Q-switched ND-YAG Laser With Topical Carbon Versus Fractional CO2 Laser for Enlarged Facial Pores
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Saadi, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: las49
Record Dates: First submitted 2020-07-04; First posted 2020-07-14 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Skin Lesion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- short pulse and Q-switched ND-YAG laser with topical carbon (Active Comparator)
  Interventions: Device: short pulse and Q-switched ND-YAG laser with topical carbon
- Fractional CO2 Laser (Active Comparator)
  Interventions: Device: fractional CO2 laser

INTERVENTIONS:
Device: short pulse and Q-switched ND-YAG laser with topical carbon — application of topical carbon cream, followed by two passes of short pulse 1064 ND-YAG, then one pass of Q-switched 1064 ND-YAG on one side of the face
  Arms: short pulse and Q-switched ND-YAG laser with topical carbon
Device: fractional CO2 laser — single pass of fractional CO2 laser on the other side of the face
  Arms: Fractional CO2 Laser

SUMMARY:
Facial pores are visible topographic features of the skin that reflect openings of pilosebaceous follicles, that may be enlarged causing distress to some individuals. Many patients desire treatment for this condition, which can be an early sign of skin aging. Therapeutic modalities include intense pulsed light, radiofrequency, dermabrasion, oral and topical retinoids, as well as chemical peeling. Lasers, as fractional CO2, short pulse and Q-switched Nd-YAG, can potentially be used in treatment of wide pores.

This study aims at the assessment and comparison of therapy with short pulsed and Q-switched Nd-YAG laser plus topical carbon with fractional CO2 laser in the management of wide facial pores.

DETAILED DESCRIPTION:
topical carbon cream will be applied to one side of the face in patients with wide facial pores, followed by 2 passes of short pulse 1064 ND:YAG laser, then one pass of Q-switched ND-YAG laser.

fractional CO2 laser will be performed to the other half of the face. the patients will receive 2 treatment sessions

ELIGIBILITY:
Inclusion Criteria:

* Participants who are more than 18 years old with the large facial pores and are aware of their problem and seeking treatment

Exclusion Criteria:

* • Previous laser therapy, chemical peeling, microdermabrasion or cosmetic procedure for the face.

  * Patients with any contraindication to laser therapy such as photosensitive diseases, skin malignancies, patients on oral retinoids.
  * Keloid-forming tendency.
  * Local or systemic treatment for skin pores in the previous 3 months
  * Connective tissue disease or the use of immunosuppressive medications.
  * Pregnancy.
  * Present or past history of herpes labialis.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-19 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2020-10-12 (Actual)

PRIMARY OUTCOMES:
the percentage of decrease in size of enlarged facial pores assessed clinically and by dermoscopy | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No